CLINICAL TRIAL: NCT07338747
Title: Does an Educational Video Increase Trial of Labor After Cesarean and Reduce Anxiety Among Women With a Prior Cesarean? A Randomized Controlled Trial
Brief Title: Educational Video, Anxiety, and Mode of Delivery After Previous Cesarean
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Wolfson Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: WOMC-0175-25
Record Dates: First submitted 2026-01-01; First posted 2026-01-14 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Anxiety; TOLAC; Previous Cesarean Delivery; Trial of Labor After Cesarean
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: Evaluation of the effect of video-based patient education on maternal anxiety levels prior to trial of labor after cesarean.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental: Video-Based Patient Education (Experimental): Participants receive structured video-based education regarding trial of labor after cesarean.
  Interventions: Behavioral: Video-Based Educational Intervention
- Active Comparator: Standard Verbal Counseling (Active Comparator): Participants receive standard verbal counseling regarding trial of labor after cesarean.
  Interventions: Other: Standard Verbal Counseling

INTERVENTIONS:
Behavioral: Video-Based Educational Intervention — A structured educational video providing information on benefits, risks, and expectations of trial of labor after cesarean.
  Arms: Experimental: Video-Based Patient Education
Other: Standard Verbal Counseling — Routine verbal counseling provided by the treating clinician regarding trial of labor after cesarean.
  Arms: Active Comparator: Standard Verbal Counseling

SUMMARY:
This interventional study evaluates whether video-based patient education regarding Trial of Labor After Cesarean (TOLAC) reduces maternal anxiety compared with standard verbal counseling. Pregnant women eligible for TOLAC will be randomized to receive either a structured educational video or routine verbal counseling. Maternal anxiety levels will be assessed using the State-Trait Anxiety Inventory (STAI).

DETAILED DESCRIPTION:
Trial of labor after cesarean (TOLAC) is a complex clinical decision that may be associated with significant maternal anxiety. Adequate counseling is essential to support informed decision-making; however, the optimal method for delivering information remains unclear.

This randomized interventional study aims to assess whether video-based patient education can reduce anxiety levels compared with standard verbal counseling. Eligible pregnant women planning delivery after a previous cesarean section will be randomly assigned to one of two study arms: video-based educational counseling or standard verbal counseling.

Anxiety will be measured using the validated State-Trait Anxiety Inventory (STAI) questionnaire after counseling. The results of this study may inform future strategies for patient counseling and shared decision-making in women considering TOLAC.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women with a singleton pregnancy.
* History of one previous cesarean delivery with a low transverse uterine incision.
* Eligible for a trial of labor after cesarean (TOLAC) according to clinical assessment and Israeli national clinical guidelines.
* Age 18 years or older.
* Hebrew-speaking.
* Ability and willingness to provide written informed consent.

Exclusion Criteria:

* Medical or obstetric conditions contraindicating vaginal delivery, including but not limited to placenta previa or marginal placenta previa.
* History of uterine surgery other than one prior low transverse cesarean section that precludes vaginal delivery.
* History of two or more prior cesarean deliveries.
* Non-vertex fetal presentation or any presentation unsuitable for a trial of labor.
* Multiple gestation.
* Diagnosed severe anxiety disorder or other significant psychiatric disorder that may interfere with participation in the study or completion of questionnaires.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Maternal Anxiety Level | Immediately after completion of counseling.
  Assessment of maternal anxiety using the State-Trait Anxiety Inventory (STAI) questionnaire.

SECONDARY OUTCOMES:
Patient Knowledge Regarding Trial of Labor After Cesarean | Immediately after completion of counseling.
  Assessment of patient knowledge regarding trial of labor after cesarean, based on a structured questionnaire developed for the study.
Rate of Successful Trial of Labor After Cesarean (TOLAC) | From delivery.
  Proportion of participants who achieved a successful vaginal birth following a trial of labor after cesarean.
Patient Satisfaction With Counseling Method | Immediately after completion of counseling.
  Patient-reported satisfaction with the counseling method received (video-based education or standard verbal counseling), assessed using a Likert-scale questionnaire.
Maternal Preference for Trial of Labor After Cesarean Versus Elective Repeat Cesarean Delivery | Immediately after completion of counseling.
  Participant-reported preference for mode of delivery (trial of labor after cesarean versus elective repeat cesarean delivery) following counseling.

CONTACTS AND LOCATIONS:
Overall Officials: Shir Lev, MD, Principal Investigator — Wolfson Medical Center

IPD SHARING:
Plan to Share IPD: No